CLINICAL TRIAL: NCT03388073
Title: Evaluation of Plant-based Nutritional Products on Stem Cells
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Natural Immune Systems Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: NIS135002
Record Dates: First submitted 2017-12-23; First posted 2018-01-02 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-02

CONDITIONS: Stem Cell Mobilization; Hematopoietic Stem Cell Mobilization; Stem Cell Homing

STUDY DESIGN:
Intervention Model Description: The study uses a randomized double-blinded placebo-controlled cross-over study design.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Both the study participants and the research staff interacting with study participants will be blinded to the plant based extract versus placebo.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Berry extract I (Experimental): Plant-based antioxidant-rich berry-based extract.
  Interventions: Other: Berry extract I
- Berry extract II (Experimental): Plant-based antioxidant-rich berry-based extract.
  Interventions: Other: Berry Extract II
- Berry extract blend (Experimental): Blend of plant-based antioxidant-rich berry-based extracts.
  Interventions: Other: Berry extract blend
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Berry extract I — Seabuckthorn berry proanthocyanidin extract 250 mg single dose
  Arms: Berry extract I
Other: Berry Extract II — Seabuckthorn berry proanthocyanidin extract 500 mg single dose
  Arms: Berry extract II
Other: Berry extract blend — Seabuckthorn berry blend with other berry-based antioxidants
  Arms: Berry extract blend
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this clinical study is to evaluate acute effects of plant-based nutritional extracts on adult stem cells, using a randomized double-blinded placebo-controlled cross-over study design.

DETAILED DESCRIPTION:
The purpose of this clinical study is to evaluate acute effects of plant-based nutritional extracts on adult stem cells, using a randomized double-blinded placebo-controlled cross-over study design. The research involves testing of acute effects of single doses of antioxidant-rich berry-based extracts, compared to a placebo. Blood samples are taken at baseline and 1 and 2 hours after consuming a single dose. The blood will be used to measure the numbers of different types of stem cells, to evaluate potential effects of stem cell mobilization and homing after consuming plant-based extracts. Adult stem cells are a type of cells that play a role in repairing and rejuvenating various tissue and organs in the body. At NIS Labs, we have shown that many types of plant-based nutritional products have small but reproducible and significant effects on stem cells, cytokines, and regenerative growth factors.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 20-75 years of age;
* Body weight higher than 110 pounds;
* BMI below 35;

Exclusion Criteria:

* Previous major gastrointestinal surgery (absorption of test product may be altered) (minor surgery not a problem);
* Currently taking daily OTC medications, such as NSAIDs, Tylenol, allergy medications, and others (birth control and 81 mg aspirin not a problem);
* Taking medications that affect the mind (such as anti-depressants) or nervous system (such as gabapentin);
* Currently experiencing intense stressful events and life changes;
* Actively depressed;
* Experiencing sleep disturbances;
* Working night shift;
* Pregnant, nursing, or trying to become pregnant;
* Food intolerances or allergies currently causing discomfort (such as Celiac's disease), due to ongoing inflammatory reactions that may negatively affect product absorption within the 3 hours of testing;
* Food allergies related to ingredients in test product.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-01-30 (Actual); Primary Completion 2019-12-20 (Estimated); Study Completion 2020-02-02 (Estimated)

PRIMARY OUTCOMES:
Change to stem cell numbers in blood circulation. | Changes at 1 and 2 hours after consumption.
  Flow cytometry evaluation of stem cell phenotype.

SECONDARY OUTCOMES:
Change to numbers of circulating CD45dim CD34+ stem cells in blood circulation. | Changes at 1 and 2 hours after consumption.
  Flow cytometry evaluation of stem cell phenotype.
Change to numbers of circulating CD45dim CD34+ CD309- stem cells in blood circulation. | Changes at 1 and 2 hours after consumption.
  Flow cytometry evaluation of stem cell phenotype.
Change to numbers of circulating CD45dim CD34+ CD309+ stem cells in blood circulation. | Changes at 1 and 2 hours after consumption.
  Flow cytometry evaluation of stem cell phenotype.
Change to numbers of circulating CD45- CD31+ CD309+ stem cells in blood circulation. | Changes at 1 and 2 hours after consumption.
  Flow cytometry evaluation of stem cell phenotype.
Change to numbers of circulating CD45- CD90+ stem cells in blood circulation. | Changes at 1 and 2 hours after consumption.
  Flow cytometry evaluation of stem cell phenotype.

CONTACTS AND LOCATIONS:
Overall Officials: Gitte Jensen, Study Director — NIS Labs
Locations (1):
- Natural Immune Systems, Klamath Falls, Oregon, United States

IPD SHARING:
Plan to Share IPD: No